CLINICAL TRIAL: NCT04392479
Title: TWICE-IRI: Optimization of Second-line Therapy With Aflibercept, Irinotecan (Day 1 or Day 1,3), 5-Fluorouracile and Folinic Acid in Patients With Metastatic Colorectal Cancer. A Randomized Phase III Study.
Acronym: TWICE-IRI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hôpital Franco-Britannique-Fondation Cognacq-Jay (Other)
Collaborators: Fondation ARCAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FBH-002
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cancer Colorectal; Metastasis
Keywords: Aflibercept
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aflibercept-FOLFIRI (arm 1) (Active Comparator): * Aflibercept (D1) H0: 4mg/kg IV infusion over 60min (+ 2-minute window),
  * Folinic acid (D1) H+1: 400mg/m² IV infusion over 120min (+ 2-minute window),
  * Irinotecan (D1) H+1: 180mg/m² IV infusion over 60min (+ 2-minute window),
  * 5-fluorouracile (D1) H+3: 400mg/m² IV infusion over 15min (+ 2-minute window),
  * 5-fluorouracile (D1 to D3): H+3.5: 2400mg/m² IV infusion over 46 hours (+ 1hour window)
  * H+49.5: End of treatment administration
  Interventions: Drug: Aflibercept-FOLFIRI
- Aflibercept-mFOLFIRI3 (arm 2) (Experimental): * Aflibercept (D1) H0: 4mg/kg IV infusion over 60min (+ 2-minute window),
  * Folinic acid (D1) H+1: 400mg/m² IV infusion over 120min (+ 2-minute window),
  * Irinotecan (D1 and D3) H+1 and H+49: 75mg/m² IV infusion over 60min (+ 2-minute window) on cycles 1 and 2, then 90mg/m² at cycle 3 and furthers in absence of AEs grade ≥2,
  * 5-fluorouracile (D1 to D3) H+3: 2400mg/m² IV infusion over 46 hours (+ 1hour window)
  * H+50: End of treatment administration
  Interventions: Drug: Aflibercept-mFOLFIRI3

INTERVENTIONS:
Drug: Aflibercept-FOLFIRI — Aflibercept-FOLFIRI
  Other Names: ZALTRAP-FOLFIRI
  Arms: Aflibercept-FOLFIRI (arm 1)
Drug: Aflibercept-mFOLFIRI3 — Aflibercept-mFOLFIRI3
  Other Names: ZALTRAP- mFOLFIRI3
  Arms: Aflibercept-mFOLFIRI3 (arm 2)

SUMMARY:
Optimization of second-line therapy with aflibercept, irinotecan (day1 or day 1,3), 5fluorouracile and folinic acid in patients with metastatic colorectal cancer. A randomized Phase III study.

DETAILED DESCRIPTION:
Background - Rationale Aflibercept The addition of aflibercept to the standard FOLFIRI regimen as second-line therapy was evaluated in a large phase III study (EFC10262-VELOUR). This combination significantly improved both PFS (4.7 to 6.9 months, HR=0.76; P=<0.001) and OS (12.1 to 13.5 months, HR=0.82; P=0.003). In the evaluable population (86.5%), the tumor response rate was also improved when adding aflibercept (ORR=19.8% [16.4-23.2]) to the FOLFIRI regimen (ORR=11.1% [8.5-13.8]).

Irinotecan The combination of aflibercept with FOLFIRI3, an optimized irinotecan-based regimen, was evaluated in 65 patients in a French multicentric retrospective cohort. (Carola C et al, WJCO 2018) In the cohort of irinotecan-naïve patients (n=30), the objective response rate was 43.3%, and the disease control rate 76.7%. Median PFS and OS were 11.3 months (95% CI 6.1-29.0) and 17.0 months (95% CI 13.0-17.3). The most common (>5%) grade 3-4 adverse events were diarrhea (37.9%), neutropenia (14.3%), stomatitis and anemia (10.4%), hypertension (6.7%).

In the cohort of patients previously treated with irinotecan (n=35), the objective response rate was 34.3%, and the disease control rate 60.0%. Median PFS and OS were 5.7 months (95% CI 3.9-10.4) and 14.3 months (95% CI 12.8-19.5).

Table. FOLFIRI-aflibercept vs. FOLFIRI3-aflibercept: a cross-trial comparison FOLFIRI-aflibercept (VELOUR) FOLFIRI3-aflibercept (Irinotecan-naïve) N = 612 N = 30 Efficacy RR, % 19.3 vs 43.3 PFS, months 6.9 vs 11.3 OS, months 13.5 vs 17.0 Grade 3-4 AEs, % Any 83.4 vs 56.7 Neutropenia 36.7 vs 14.3 Diarrhea 19.3 vs 37.9 Mucositis 13.8 vs 10.4 Hypertension 19.3 vs 6.9 Discontinuation, % Progression 49.8 vs 36.7 Adverse event 26.6 vs 46.7

Study Objectives

Primary:

•To compare once (day 1) or twice (day 1, day 3) administration of irinotecan in combination with 5-fluorouracile and aflibercept as second-line therapy in patients with metastatic colorectal cancer in terms of overall response rate (ORR)

Secondary:

* To evaluate disease control rate (DRC) and Early Response Rate (ERR)
* To evaluate progression-free survival (PFS) and overall survival (OS),
* to evaluate the conversion rate to locoregional therapy, surgery of metastasis, the quality of resection (R0, R1, R2) and the pathological response in patients with resected metastatic disease,
* To assess the impact on health-related quality of life (HRQOL) using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-C30 (QLQ-C30),
* To assess Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) on using the National Cancer Institute Common Toxicity Criteria (NCI-CTC version 5.0).

Exploratory:

* To assess the impact on selected circulating biomarkers (angiogenic and exosomal)
* To assess the impact on selected tumor biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent and stated willingness to comply with all study procedures and availability for the duration of the study, Signed, written Informed Consent Form (ICF),
2. Willing and able to comply with the protocol,
3. Age 18-75 years,
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1,
5. Life expectancy ≥ 3 months,
6. Histologically proven carcinoma of colon and/or rectum,
7. Confirmed unresectable metastatic disease,
8. At least one measurable and/or evaluable tumor metastasis on CT-scan or MRI per RECIST criteria version 1.1,
9. Prior oxaliplatin-based first-line therapy for metastatic disease (the use of prior bevacizumab or anti-EGFR mabs is allowed but not mandatory) - Less than 6 months from completion of any prior oxaliplatin-based adjuvant therapy can be considered as first-line therapy. Prior use of irinotecan in combination with oxaliplatin and 5FU as first-line therapy is allowed if the interval between the last administration of irinotecan and disease progression is at least 6 months (ie, irinotecan-free interval ≥6 months).
10. Negative urine and/or serum pregnancy test within 7 days before inclusion if female subject is of childbearing potential,
11. Clinical laboratory parameters adequate as follows:

    * Serum total bilirubin level ≤ 1.5 x upper normal limit (UNL),
    * Neutrophil count ≥ 1.5x109/L,
    * Platelet count ≥ 100x109/L,
    * Hemoglobin ≥ 9 g/dL,
    * Serum creatinine level ≤ 150µM,
    * Serum albumin ≥ 25 g/L,
    * Calcium ≥ 1 x ULN
    * Alkaline phosphatase (ALP) < 3 x ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN (in the case of liver metastases, <5 x ULN),
    * Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour,
12. For women of childbearing potential and for men, agreement to use an effective contraceptive method from the time of screening throughout the study until 6 months after administration of the last dose of any study medication. Highly effective contraceptive method consist of prior sterilization, inter-uterine device, intrauterine hormone-releasing system, oral or injectable contraceptives barrier methods, and/or true sexual abstinence),
13. Affiliation to French health care system.

Exclusion Criteria:

1. History of arterial thrombotic event in the last 6 months (eg., myocardial infarction, cerebrovascular accident or transient ischemic attack),
2. Uncontrolled hypertension (defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg despite optimal medical therapy), or history of hypertensive crisis, or hypertensive encephalopathy,
3. Prior use of aflibercept,
4. Adverse events from prior anticancer therapy grade ≥2 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0), except for neuropathy and alopecia,
5. Bowel obstruction, inflammatory bowel disease
6. Known DPD deficiency. If not known for the patient, testing for DPD should be done during the screening period (patients with uracilemia ≥16ng/mL are not eligible),
7. Known UGT1A1 deficiency (eg, Gilbert syndrome, Crigler-Najjar syndrome). If not known for the patient, genetic testing for UGT1A1 should be done during the screening period for patients with hyperbilirubinemia (ie, total bilirubin level >1xULN),
8. Active infection requiring intravenous antibiotics at the start of study treatment,
9. Known active infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV),
10. Known allergy or hypersensitivity to the active substance or ingredients of any study drug,
11. Women currently pregnant or breastfeeding,
12. Inability to comply with study and follow-up procedures as judged by the Investigator,
13. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy)
14. Concomitant use of Saint John Wort herb (millepertuis), Yellow Fever vaccine, Live Attenuated Vaccines (LAV) and phenytoine
15. Treatment with any other investigational medicinal product within 28 days or 5 investigational agent half-lives (whichever is longer) prior to the start of study treatment,
16. Any other disease, active, uncontrolled bacterial, viral or fungal infection requiring systemic therapy, metabolic dysfunction, physical examination finding or clinical laboratory finding that leads to reasonable suspicion of a disease or condition that contraindicates the use of study drugs that may affect the interpretation of the results, or that may render the subject at high risk for treatment complications.
17. Previous or concurrent malignancy, except for adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for three years prior to study entry,
18. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to start of study treatment, or anticipation of need for major surgical procedure during the course of the study.
19. Minor surgical procedure including placement of a vascular access device, within 2 days of start of study treatment,
20. History of abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to start study treatment.
21. Clinically significant active cardiac disease (including NYHA class III or IV congestive heart failure)
22. Venous thromboembolic event (including pulmonary embolism) grade 3 or 4 within 6 months prior to start study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR). | 2 months
  Tumor measurements will be obtained using CT-scans (or MRIs) of the thorax, abdomen, and pelvis at baseline then every 8 weeks (+/- one week) according to RECIST v1.1. At the investigator's discretion, tumor assessments may be repeated at any time if progressive disease is suspected.
  It is preferred that the scans for a patient are taken with the same technique (CT or MRI) throughout the study.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 2 months
  The disease control rate is the sum of patients with tumor response (either CR or PR) or stabilization (SD) as best response.
Early response rate | 2 months
  The early response rate will be evaluated at the first tumor evaluation at 8 weeks (+/- 1 week).
Progression-free survival (PFS) | 2 months
  PFS is defined as the time interval from randomization to the date of first documented disease progression or death from any cause, whichever occurs first. Alive patients without progression will be censored at the last tumor assessment, either during study treatment period or during follow-up period.
Overall survival (OS) | time interval from randomization to the date of death from any cause. Assessed up to 13 months after the beginning of the study
  OS is defined as the time interval from randomization to the date of death from any cause. Alive patients will be censored at the last date known to be alive, either during study treatment period or during follow-up period. Survival status will be assessed by telephone, ordinary visits, hospital records or other means found suitable until death or the end of the study, whichever occurs first. Information regarding post-study anti-cancer therapies will be collected if new treatment is initiated.
Salvage surgery rate | 2 months
  Salvage surgery rate (%) corresponding to the number of patients amenable to surgery of metastasis during study treatment. The number of patients with R0 or R1 resection will be evaluated.
Pathological response rate | 2 months
  The pathological tumor response will be assessed in patients having primary and/or metastasis resection using Tumor Regression Grade (TRG), modified TRG and Blazer grade. (Rubbia-Brandt L et al, Ann Oncol 2007 ; Blazer 3rd DG et al, J Clin Oncol 2008)
Tolerance | 2 weeks
  frequency of AEs and SAEs per patient and per cycle of treatment using NCI CTCAE v5.0.
HRQoL | 2 months
  The time until definitive HRQoL score deterioration (TUDD), (Bonnetain F et al, Eur J Cancer 2010) The survival without HRQoL deterioration-free survival (QFS). HRQoL will be assessed with EORTC QLQ-C30 questionnaire
Exploratory biomarkers | 2 months
  Blood : (PlGF, VEGF-A, VEGF-B, VEGF-C, VEGF-D, sVEGFR1, sVEGFR2, sVEGFR3, Ang2, sTie2, Syndecan) .Exosomal biomarkers assessments (CEA, HSP70, VEGFR-2)
  Tumor: Analyses will be performed according to the knowledge on potential markers at that time

CONTACTS AND LOCATIONS:
Overall Officials: Benoist CHIBAUDEL, MD, Principal Investigator — Franco-British Hospital GCS IHFB Cognacq-Jay
Locations (1):
- Franco-British Hospital - GCS IHFB Cognacq-Jay, Levallois-Perret, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Tournigand C, Andre T, Achille E, Lledo G, Flesh M, Mery-Mignard D, Quinaux E, Couteau C, Buyse M, Ganem G, Landi B, Colin P, Louvet C, de Gramont A. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004 Jan 15;22(2):229-37. doi: 10.1200/JCO.2004.05.113. Epub 2003 Dec 2. PMID 14657227
- [Background] Jolivet J. Role of leucovorin dosing and administration schedule. Eur J Cancer. 1995 Jul-Aug;31A(7-8):1311-5. doi: 10.1016/0959-8049(95)00140-e. PMID 7577042
- [Background] Van Cutsem E, Tabernero J, Lakomy R, Prenen H, Prausova J, Macarulla T, Ruff P, van Hazel GA, Moiseyenko V, Ferry D, McKendrick J, Polikoff J, Tellier A, Castan R, Allegra C. Addition of aflibercept to fluorouracil, leucovorin, and irinotecan improves survival in a phase III randomized trial in patients with metastatic colorectal cancer previously treated with an oxaliplatin-based regimen. J Clin Oncol. 2012 Oct 1;30(28):3499-506. doi: 10.1200/JCO.2012.42.8201. Epub 2012 Sep 4. PMID 22949147
- [Background] Peeters M, Price TJ, Cervantes A, Sobrero AF, Ducreux M, Hotko Y, Andre T, Chan E, Lordick F, Punt CJ, Strickland AH, Wilson G, Ciuleanu TE, Roman L, Van Cutsem E, Tzekova V, Collins S, Oliner KS, Rong A, Gansert J. Randomized phase III study of panitumumab with fluorouracil, leucovorin, and irinotecan (FOLFIRI) compared with FOLFIRI alone as second-line treatment in patients with metastatic colorectal cancer. J Clin Oncol. 2010 Nov 1;28(31):4706-13. doi: 10.1200/JCO.2009.27.6055. Epub 2010 Oct 4. PMID 20921462
- [Background] Tabernero J, Yoshino T, Cohn AL, Obermannova R, Bodoky G, Garcia-Carbonero R, Ciuleanu TE, Portnoy DC, Van Cutsem E, Grothey A, Prausova J, Garcia-Alfonso P, Yamazaki K, Clingan PR, Lonardi S, Kim TW, Simms L, Chang SC, Nasroulah F; RAISE Study Investigators. Ramucirumab versus placebo in combination with second-line FOLFIRI in patients with metastatic colorectal carcinoma that progressed during or after first-line therapy with bevacizumab, oxaliplatin, and a fluoropyrimidine (RAISE): a randomised, double-blind, multicentre, phase 3 study. Lancet Oncol. 2015 May;16(5):499-508. doi: 10.1016/S1470-2045(15)70127-0. Epub 2015 Apr 12. PMID 25877855
- [Background] Guichard S, Cussac D, Hennebelle I, Bugat R, Canal P. Sequence-dependent activity of the irinotecan-5FU combination in human colon-cancer model HT-29 in vitro and in vivo. Int J Cancer. 1997 Nov 27;73(5):729-34. doi: 10.1002/(sici)1097-0215(19971127)73:53.0.co;2-#. PMID 9398054
- [Background] Mullany S, Svingen PA, Kaufmann SH, Erlichman C. Effect of adding the topoisomerase I poison 7-ethyl-10-hydroxycamptothecin (SN-38) to 5-fluorouracil and folinic acid in HCT-8 cells: elevated dTTP pools and enhanced cytotoxicity. Cancer Chemother Pharmacol. 1998;42(5):391-9. doi: 10.1007/s002800050835. PMID 9771954
- [Background] Mans DR, Grivicich I, Peters GJ, Schwartsmann G. Sequence-dependent growth inhibition and DNA damage formation by the irinotecan-5-fluorouracil combination in human colon carcinoma cell lines. Eur J Cancer. 1999 Dec;35(13):1851-61. doi: 10.1016/s0959-8049(99)00222-1. PMID 10674003
- [Background] Falcone A, Di Paolo A, Masi G, Allegrini G, Danesi R, Lencioni M, Pfanner E, Comis S, Del Tacca M, Conte P. Sequence effect of irinotecan and fluorouracil treatment on pharmacokinetics and toxicity in chemotherapy-naive metastatic colorectal cancer patients. J Clin Oncol. 2001 Aug 1;19(15):3456-62. doi: 10.1200/JCO.2001.19.15.3456. PMID 11481350
- [Background] Mabro M, Louvet C, Andre T, Carola E, Gilles-Amar V, Artru P, Krulik M, de Gramont A; GERCOR. Bimonthly leucovorin, infusion 5-fluorouracil, hydroxyurea, and irinotecan (FOLFIRI-2) for pretreated metastatic colorectal cancer. Am J Clin Oncol. 2003 Jun;26(3):254-8. doi: 10.1097/01.COC.0000020581.59835.7A. PMID 12796595
- [Background] Mabro M, Artru P, Andre T, Flesch M, Maindrault-Goebel F, Landi B, Lledo G, Plantade A, Louvet C, de Gramont A. A phase II study of FOLFIRI-3 (double infusion of irinotecan combined with LV5FU) after FOLFOX in advanced colorectal cancer patients. Br J Cancer. 2006 May 8;94(9):1287-92. doi: 10.1038/sj.bjc.6603095. PMID 16622455
- [Background] Bidard FC, Tournigand C, Andre T, Mabro M, Figer A, Cervantes A, Lledo G, Bengrine-Lefevre L, Maindrault-Goebel F, Louvet C, de Gramont A. Efficacy of FOLFIRI-3 (irinotecan D1,D3 combined with LV5-FU) or other irinotecan-based regimens in oxaliplatin-pretreated metastatic colorectal cancer in the GERCOR OPTIMOX1 study. Ann Oncol. 2009 Jun;20(6):1042-7. doi: 10.1093/annonc/mdn730. Epub 2009 Jan 19. PMID 19153116
- [Background] Chibaudel B, Maindrault-Goebel F, Bachet JB, Louvet C, Khalil A, Dupuis O, Hammel P, Garcia ML, Bennamoun M, Brusquant D, Tournigand C, Andre T, Arbaud C, Larsen AK, Wang YW, Yeh CG, Bonnetain F, de Gramont A. PEPCOL: a GERCOR randomized phase II study of nanoliposomal irinotecan PEP02 (MM-398) or irinotecan with leucovorin/5-fluorouracil as second-line therapy in metastatic colorectal cancer. Cancer Med. 2016 Apr;5(4):676-83. doi: 10.1002/cam4.635. Epub 2016 Jan 24. PMID 26806397
- [Background] Carola C, Ghiringhelli F, Kim S, Andre T, Barlet J, Bengrine-Lefevre L, Marijon H, Garcia-Larnicol ML, Borg C, Dainese L, Steuer N, Richa H, Benetkiewicz M, Larsen AK, de Gramont A, Chibaudel B. FOLFIRI3-aflibercept in previously treated patients with metastatic colorectal cancer. World J Clin Oncol. 2018 Sep 14;9(5):110-118. doi: 10.5306/wjco.v9.i5.110. PMID 30254966
- [Background] Ghiringhelli F, Vincent J, Beltjens F, Bengrine L, Ladoire S. Fluorouracil, leucovorin and irinotecan associated with aflibercept can induce microscopic colitis in metastatic colorectal cancer patients. Invest New Drugs. 2015 Dec;33(6):1263-6. doi: 10.1007/s10637-015-0295-6. Epub 2015 Oct 22. PMID 26490656
- [Background] Rubbia-Brandt L, Giostra E, Brezault C, Roth AD, Andres A, Audard V, Sartoretti P, Dousset B, Majno PE, Soubrane O, Chaussade S, Mentha G, Terris B. Importance of histological tumor response assessment in predicting the outcome in patients with colorectal liver metastases treated with neo-adjuvant chemotherapy followed by liver surgery. Ann Oncol. 2007 Feb;18(2):299-304. doi: 10.1093/annonc/mdl386. Epub 2006 Oct 23. PMID 17060484
- [Background] Blazer DG 3rd, Kishi Y, Maru DM, Kopetz S, Chun YS, Overman MJ, Fogelman D, Eng C, Chang DZ, Wang H, Zorzi D, Ribero D, Ellis LM, Glover KY, Wolff RA, Curley SA, Abdalla EK, Vauthey JN. Pathologic response to preoperative chemotherapy: a new outcome end point after resection of hepatic colorectal metastases. J Clin Oncol. 2008 Nov 20;26(33):5344-51. doi: 10.1200/JCO.2008.17.5299. Epub 2008 Oct 20. PMID 18936472
- [Background] Bonnetain F, Dahan L, Maillard E, Ychou M, Mitry E, Hammel P, Legoux JL, Rougier P, Bedenne L, Seitz JF. Time until definitive quality of life score deterioration as a means of longitudinal analysis for treatment trials in patients with metastatic pancreatic adenocarcinoma. Eur J Cancer. 2010 Oct;46(15):2753-62. doi: 10.1016/j.ejca.2010.07.023. Epub 2010 Aug 17. PMID 20724140